CLINICAL TRIAL: NCT04757974
Title: A Two-Part Randomized Study to Evaluate the Relative Bioavailability of Temsavir Following Single Dose Administration of Fostemsavir 600 mg Tablets Compared to Two Fostemsavir 200 mg Tablet Formulations and to Evaluate the Effect of Food on Bioavailability of Selected Fostemsavir 200 mg Tablet Formulation in Healthy Adult Participants
Brief Title: Low-dose Fostemsavir Extended Release Relative Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 213075
Expanded Access: NCT04233047 (Available)
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: HIV Infections
Keywords: Temsavir; Fostemsavir; Bioavailability; Extended Release tablet; GSK3684934; Food effect
MeSH Terms: conditions — HIV Infections | interventions — fostemsavir

STUDY DESIGN:
Intervention Model Description: This is a two-part study, where Part 1 will be conducted as a randomized three period, three treatment crossover study and Part 2 will have a randomized two period, two treatment crossover design.
Masking Description: This is an open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1: Treatment sequence ABC (Experimental): Participants will receive FTR 3×200 mg ER tablets (Treatment A) in Period 1 followed by FTR 3×200 mg ER tablets (Treatment B) in Period 2 followed by FTR 600 mg ER tablet (Treatment C, reference) in Period 3.
  Interventions: Drug: Fostemsavir 600 mg; Drug: Fostemsavir 200 mg
- Part 1: Treatment sequence BCA (Experimental): Participants will receive FTR 3×200 mg ER tablets (Treatment B) in Period 1 followed by FTR 600 mg ER tablet (Treatment C, reference) in Period 2 followed by FTR 3×200 mg ER tablets (Treatment A) in Period 3.
  Interventions: Drug: Fostemsavir 600 mg; Drug: Fostemsavir 200 mg
- Part 1: Treatment sequence CAB (Experimental): Participants will receive FTR 600 mg ER tablet in Period 1 (Treatment C, reference) followed by FTR 3×200 mg ER tablets (Treatment A) in Period 2 followed by FTR 3×200 mg ER tablets (Treatment B) in Period 3.
  Interventions: Drug: Fostemsavir 600 mg; Drug: Fostemsavir 200 mg
- Part 1: Treatment sequence ACB (Experimental): Participants will receive FTR 3×200 mg ER tablets (Treatment A) in Period 1 followed by FTR 600 mg ER tablet (Treatment C, reference) in Period 2 followed by FTR 3×200 mg ER tablets (Treatment B) in Period 3.
  Interventions: Drug: Fostemsavir 600 mg; Drug: Fostemsavir 200 mg
- Part 1: Treatment sequence BAC (Experimental): Participants will receive FTR 3×200 mg ER tablets (Treatment B) in Period 1 followed by FTR 3×200 mg ER tablets (Treatment A) in Period 2 followed by FTR 600 mg ER tablet (Treatment C, reference) in Period 3.
  Interventions: Drug: Fostemsavir 600 mg; Drug: Fostemsavir 200 mg
- Part 1: Treatment sequence CBA (Experimental): Participants will receive FTR 600 mg ER tablet (Treatment C, reference) in Period 1 followed by FTR 3×200 mg ER tablets (Treatment B) in Period 2 followed by FTR 3×200 mg ER tablets (Treatment A) in Period 3.
  Interventions: Drug: Fostemsavir 600 mg; Drug: Fostemsavir 200 mg
- Part 2: Treatment sequence DE (Experimental): Participants will receive the selected low-dose formulation of FTR 3 × 200 mg ER tablets in a fasted state (Treatment D) in Period 1 and following a high fat high calorie meal (Treatment E) in Period 2.
  Interventions: Drug: Fostemsavir 200 mg
- Part 2: Treatment sequence ED (Experimental): Participants will receive the selected low-dose formulation of FTR 3 × 200 mg ER tablets following a high fat high calorie meal (Treatment E) in Period 1 and in a fasted state (Treatment D) in Period 2.
  Interventions: Drug: Fostemsavir 200 mg

INTERVENTIONS:
Drug: Fostemsavir 600 mg — Fostemsavir tablets will be administered via oral route.
  Arms: Part 1: Treatment sequence ABC; Part 1: Treatment sequence ACB; Part 1: Treatment sequence BAC; Part 1: Treatment sequence BCA; Part 1: Treatment sequence CAB; Part 1: Treatment sequence CBA
Drug: Fostemsavir 200 mg — Fostemsavir tablets will be administered via oral route.

SUMMARY:
This is a two-part study. Part 1 will evaluate relative bioavailability of temsavir (TMR) following single dose administration of the reference fostemsavir (FTR) compared to two low-dose ER tablet formulations of FTR. In Part 2, the effect of food on the bioavailability of TMR will be assessed on the selected low-dose ER tablet formulation from Part 1.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age inclusive.
* Healthy as determined by the investigator or medically qualified designee.
* A participant with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator, in consultation with the Medical Monitor, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 kilograms (kg) (110 pounds [lbs.]) for men and >= 45 kg (99 lbs.) for women and body mass index (BMI) within the range 18.5-31.0 kilogram per meter square (kg/m^2) (inclusive).
* Male participants are eligible to participate if they agree to use contraceptive methods.
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies: Is a woman of non-childbearing potential (WONCBP). OR Is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Alanine transaminase (ALT) >1.5x upper limit of normal (ULN).
* Total bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if total bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 millisecond (msec) for males and QTcF>470 msec for females.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and ViiV/GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise participant safety.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliters (mL) within 56 days.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrollment or past participation within the last 30 days or five half-lives whichever is longer, before signing of consent in any other clinical study involving an investigational study intervention or any other type of medical research.
* Presence of hepatitis B surface antigen (HBsAg) [or hepatitis B core antibody (HBcAb)] at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C Ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention.
* Positive Human immunodeficiency virus (HIV)-1 and -2 antigen/antibody immunoassay.
* Cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females.
* Regular use of known drugs of abuse.
* Sensitivity to heparin or heparin-induced thrombocytopenia.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* A participant with a history of beta-lactam allergy, regardless of severity/seriousness.
* A participant with known or suspected active Coronavirus disease-2019 (COVID-19) infection OR contact with an individual with known COVID-19, within 14 days of study enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Part 1: Area under the plasma concentration-time curve (AUC) from time zero to the last quantifiable time point (AUC[0-t]) of temsavir | Predose (Day 1) until 72 hour post dose
Part 1: AUC from time zero extrapolated to infinite time (AUC[0-infinity]) of temsavir | Predose (Day 1) until 72 hour post dose
Part 1: Maximum observed plasma concentration (Cmax) | Predose (Day 1) until 72 hour post dose

SECONDARY OUTCOMES:
Part 1: Time to Cmax (Tmax) of temsavir | Predose (Day 1) until 72 hour post dose
Part 1: Elimination half-life (T1/2) of temsavir | Predose (Day 1) until 72 hour post dose
Part 1: Concentration at 12 hours post-dose of temsavir | 12 hours post-dose
Part 1 and Part 2: Number of participants with clinically significant change from Baseline in vital signs and clinical laboratory parameters | Baseline (Day -1) until end of follow up at 4 weeks
Part 1 and Part 2: Number of participants reporting adverse events (AEs) and serious adverse events (SAEs) | Baseline (Day -1) until end of follow up at 4 weeks
Part 2: AUC [0-t] of temsavir | Predose (Day 1) until 72 hour post dose
Part 2: AUC [0-infinity] of temsavir | Predose (Day 1) until 72 hour post dose
Part 2: Cmax of temsavir | Predose (Day 1) until 72 hour post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.